CLINICAL TRIAL: NCT01258777
Title: A Phase I Study to Evaluate the Safety and Pharmacokinetics of CNTO 148 Following Single Subcutaneous Administration to Healthy Japanese and Caucasian Subjects
Brief Title: A Study of the Pharmacokinetics of Golimumab in Japanese and Caucasian Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR016345
Record Dates: First submitted 2010-11-22; First posted 2010-12-13 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Japanese male; Caucasian male; Simponi
MeSH Terms: interventions — golimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): 200 mg golimumab or placebo Single dose of 200 mg subcutaneously
  Interventions: Drug: 200 mg golimumab or placebo
- 002 (Experimental): 400 mg golimumab or placebo Single dose of 400 mg subcutaneously
  Interventions: Drug: 400 mg golimumab or placebo

INTERVENTIONS:
Drug: 400 mg golimumab or placebo — Single dose of 400 mg subcutaneously
  Arms: 002
Drug: 200 mg golimumab or placebo — Single dose of 200 mg subcutaneously
  Arms: 001

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics of golimumab in Japanese and Caucasian Males.

DETAILED DESCRIPTION:
This is a randomized (study medication assigned by chance), double-blind (both the physician and subject do not know the assigned study medication) study to assess the safety, tolerability, immune response, pharmacokinetics (what the body does to the drug), of golimumab (Simponi). The study population will consist of 24 healthy male Japanese subjects and 24 healthy male Caucasian subjects. Subjects will receive a single dose of either 200 mg or 400 mg golimumab or placebo. Subjects will be in the study for up to 16 weeks. Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (eg, blood pressure), and the occurrence and severity of adverse events. A single dose of 200 mg or 400 mg golimumab, or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Have no clinically relevant abnormalities
* non-smoker or agree to smoke no more than 10 cigarettes or 2 cigars per day throughout the study
* Japanese subjects born in Japan, outside of Japan for no more than 5 years, and have Japanese parents and maternal and paternal grandparents, determined by subject's verbal report
* Japanese subjects must have a valid Japanese passport
* Caucasian subjects must have Caucasian parents.

Exclusion Criteria:

* Have or had a history of clinically significant, severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease
* Have any underlying physical or psychological medical condition
* Be unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2010-10; Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (study of what the body does to the drug) of golimumab in Japanese and Caucasian Male subjects | Week 12 (Day 78)
Determine the immune response of golimumab in Japanese and Caucasian Male subjects | Week 12 (Day 78)
Safety of golimumab in Japanese and Caucasian Male subjects | Week 12 (Day 78)
Tolerability of golimumab in Japanese and Caucasian Male subjects | Week 12 (Day 78)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (1):
- Cypress, California, United States